CLINICAL TRIAL: NCT03053336
Title: App-technology to Enhance Self-care for Patients With Diabetes Type 2 - A Randomized Controlled Trial
Brief Title: App-technology to Increase Physical Activity Among Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Ylva Trolle Lagerros, MD, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnr: 2016/2041-31/2
Record Dates: First submitted 2017-02-07; First posted 2017-02-15 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes Mellitus; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App-technology group (Experimental): Participants in the intervention group (App-technology) will use a newly developed smartphone application ("app") in which steps are automatically measured and laboratory values from blood sampling within primary care will be shown.
  Intervention: App-technology to increase physical activity
  Interventions: Behavioral: App-technology to increase physical activity
- Control group (No Intervention): The control group will receive standard care

INTERVENTIONS:
Behavioral: App-technology to increase physical activity — Access to the smartphone-app during 12 weeks. A personal step goal is set for each individual in the app.
  Arms: App-technology group

SUMMARY:
The aim of this study is to investigate the effect of using new app-based technology to improve self-care, compared to usual care in patients with type 2 diabetes. The hypothesis is that the intervention, i.e. using the new technology, will have a greater positive effect on physical activity levels and outcomes of HbA1c than usual care.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of type 2 diabetes
* 18 years of age or older
* Ability to communicate in Swedish
* Have and be able to use a smartphone

Exclusion Criteria:

* Not being able to walk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in physical activity level (counts/min from accelerometers) | baseline and month 3, 6 and 12

SECONDARY OUTCOMES:
HbA1c (mmol/mol) | Baseline and month 3, 6 and 12
Steps/day | Baseline and month 3, 6 and 12
Total cholesterol (mmol/L) | Baseline and month 3, 6 and 12
HDL-cholesterol (mmol/L) | Baseline and month 3, 6 and 12
Triglycerides (mmol/L) | Baseline and month 3, 6 and 12
Apolipoprotein A1 (g/l) | Baseline and month 3, 6 and 12
Apolipoprotein B (g/l) | Baseline and month 3, 6 and 12
Body weight (kg) | Baseline and month 3, 6 and 12
Body Mass Index (BMI, kg/m2) | Baseline and month 3, 6 and 12
Body composition | Baseline and month 3, 6 and 12
  Including: %Body Fat, Fat free mass (kg), Muscle mass (kg), Total body water (kg, %)
Waist circumference (cm) | Baseline and month 3, 6 and 12
Blood pressure (mmHg) | Baseline and month 3, 6 and 12

OTHER OUTCOMES:
Change in dietary habits assessed using a food frequency questionnaire | Baseline and month 3, 6 and 12
Change in tobacco use habits (smoking and Swedish snuff use) | Baseline and month 3, 6 and 12
Change in sleeping habits assessed using a 13 item questionnaire | Baseline and month 3, 6 and 12
Change in perceived purpose in life | Baseline and month 3, 6 and 12
Change in perceived stress levels using the perceived stress scale | Baseline and month 3, 6 and 12
Change in reported self-efficacy for exercise | Baseline and month 3, 6 and 12
  One's confidence in walking is assessed
Change in reported self-efficacy diabetes is assessed using a 20 item questionnaire | Baseline and month 3, 6 and 12
Change in RAND-36 | Baseline and month 3, 6 and 12
Change in neighborhood Environment assessed by questions on safety and walking environment | Baseline and month 3, 6 and 12
Social support for exercise assessed using a 6 item questionnaire | Baseline and month 3, 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Ylva Trolle Lagerros, MD, PhD, Principal Investigator — Karolinska Institutet and Stockholm County Councill
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonn SE, Hummel M, Peveri G, Eke H, Alexandrou C, Bellocco R, Lof M, Trolle Lagerros Y. Effectiveness of a Smartphone App to Promote Physical Activity Among Persons With Type 2 Diabetes: Randomized Controlled Trial. Interact J Med Res. 2024 Mar 21;13:e53054. doi: 10.2196/53054. PMID 38512333
- [Derived] Sjoblom L, Bonn SE, Alexandrou C, Dahlgren A, Eke H, Trolle Lagerros Y. Dietary habits after a physical activity mHealth intervention: a randomized controlled trial. BMC Nutr. 2023 Feb 2;9(1):23. doi: 10.1186/s40795-023-00682-4. PMID 36732788
- [Derived] Hummel M, Bonn SE, Trolle Lagerros Y. The effect of the smartphone app DiaCert on health related quality of life in patients with type 2 diabetes: results from a randomized controlled trial. Diabetol Metab Syndr. 2022 Dec 17;14(1):192. doi: 10.1186/s13098-022-00965-z. PMID 36528609
- [Derived] Bonn SE, Alexandrou C, Hjorleifsdottir Steiner K, Wiklander K, Ostenson CG, Lof M, Trolle Lagerros Y. App-technology to increase physical activity among patients with diabetes type 2 - the DiaCert-study, a randomized controlled trial. BMC Public Health. 2018 Jan 10;18(1):119. doi: 10.1186/s12889-018-5026-4. PMID 29316905